CLINICAL TRIAL: NCT02796131
Title: A Phase I, Single-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of Different Multiple Dose Regimens of RDX5791 in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacodynamics of RDX5791 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RDX5791-102
Record Dates: First submitted 2016-06-07; First posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: Phase I; Healthy; Pharmacodynamics
MeSH Terms: interventions — tenapanor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- 30 mg bid (Experimental): 30 mg of RDX5791 administered twice daily PO (60 mg total dose/day).
  Interventions: Drug: RDX5791; Drug: Placebo
- 30 mg tid (Experimental): 30 mg of RDX5791 administered three times daily PO (90 mg total dose/day).
  Interventions: Drug: RDX5791; Drug: Placebo
- 60 mg bid (Experimental): 60 mg of RDX5791 administered two times daily (120 mg total dose/day).
  Interventions: Drug: RDX5791; Drug: Placebo
- 15 mg bid (Experimental): 15 mg of RDX5791 administered two times daily (30 mg total dose/day).
  Interventions: Drug: RDX5791; Drug: Placebo
- 30 mg QD (Experimental): 30 mg of RDX5791 administered once daily (30 mg total dose/day).
  Interventions: Drug: RDX5791; Drug: Placebo
- Escalating dose bid (Experimental): 15 mg or 30 mg or 45 mg of RDX5791 administered two times daily (30, 60, or 90 mg total dose/day respectively). The stopping criteria for the dose escalation is based on Bristol Stool Score and AEs.
  Interventions: Drug: RDX5791; Drug: Placebo
- 30 mg bid with psyllium (Experimental): 30 mg of RDX5791 administered two times daily (60 mg total dose/day) with psyllium taken up to three times per day (maximum of 15 g psyllium/day).
  Interventions: Drug: RDX5791; Drug: Placebo

INTERVENTIONS:
Drug: RDX5791
  Other Names: Tenapanor; AZD1722
Drug: Placebo — Placebo

SUMMARY:
A Phase 1, single-center, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerabiltiy, and pharmacodynamics of different multiple dose regimens of RDX5791 in healthy volunteers.

DETAILED DESCRIPTION:
The starting doses for this study are based on the results from the multiple ascending-dose study performed on RDX5791 (Protocol RDX5791-101). Subjects will be screened within 3 weeks of check in to the CPU. Each cohort of 15 subjects (12 RDX5791, 3 placebo) will check in to the CPU on Day -5 before dinner. Each subject will receive a diet standardized for Na+ content while in the CPU. Subjects will receive doses of RDX5791 with approximately 240 mL of non-carbonated water on Days 1 to 7 (just prior to meals, depending on QD, bid, or tid regimens). Subjects will be provided standardized meals within 10 minutes after dosing. Doses can be administered with breakfast, lunch, or dinner.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 29.9 kg/m², inclusive
* No clinically significant abnormalities in medical history
* Females must be non-pregnant, non-lactating, and either postmenopausal for at least 12 months or have agreed to use an effective form of contraception from the time of signing the informed consent until 45 days after end of study
* Men must be either sterile, abstinent, or agreed to use an approved method of contraception from check-in until 45 days after final study visit

Exclusion Criteria:

* Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the GI tract
* Any surgery on the small intestine or colon, excluding appendectomy
* Loose stools (Bristol Stool Form Score of 6 or 7) ≥2 days in the past 7 days
* Hepatic dysfunction ([ALT] or [AST]) >1.5 times the upper limit of normal or renal impairment
* Any evidence of or treatment of malignancy, excluding non-melanomatous malignancies of the skin
* Use of diuretic medications, medications that are known to affect stool consistency and/or GI motility
* Use of an investigational agent within 30 days prior to Day -2
* Positive virology, alcohol, or drugs of abuse test during screening
* Use of any prescription medication within 7 days before admission to the CPU
* Have had significant blood loss (>450 mL) or have donated 1 or more units of blood or plasma within 8 weeks prior to study entry

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety of different dosing regimens of RDX5791 | 7 Days
  Safety assessments will be based on adverse events, clinical laboratory tests, vital signs, ECG, and physical exams.

SECONDARY OUTCOMES:
Pharmacodynamics of different dosing regimens of RDX5791 | 7 Days
  Pharmacodynamics of different dosing regimens of RDX5791 will be assessed by bowel movement timing, consistency, frequency, and by urine and stool sodium (Na+) excretion.

CONTACTS AND LOCATIONS:
Overall Officials: David P. Rosenbaum, Ph.D, Study Chair — Ardelyx, Inc.

REFERENCES:
- [Derived] Rosenbaum DP, Yan A, Jacobs JW. Pharmacodynamics, Safety, and Tolerability of the NHE3 Inhibitor Tenapanor: Two Trials in Healthy Volunteers. Clin Drug Investig. 2018 Apr;38(4):341-351. doi: 10.1007/s40261-017-0614-0. PMID 29363027